CLINICAL TRIAL: NCT04824027
Title: Predicting Response to Neoadjuvant Chemotherapy Using Harmonic Motion Imaging in Women With Breast Cancer
Brief Title: Breast Elasticity Imaging During Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisa Konofagou, Robert and Margaret Hariri Professor in Biomedical Engineering and Radiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT4412; R01CA228275 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; Harmonic Motion Imaging (HMI); Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMI Group (Experimental): Women undergoing standard neoadjuvant chemotherapy for breast cancer
  Interventions: Procedure: Harmonic motion imaging

INTERVENTIONS:
Procedure: Harmonic motion imaging — Harmonic motion imaging (HMI) is a non-invasive ultrasound elasticity imaging technique that yields a quantitative relative measurement of tissue stiffness suitable for comparisons between individuals and over time. This technique induces dynamic tissue vibrations internally for tissue elasticity characterization. Participants will be asked to lie down on their back, hold still with shallow breathing while pictures/images are taken of the breast where the tumor is located using an ultrasound without any invasive procedures.
  Other Names: HMI technique

SUMMARY:
For this study, the investigators propose investigation of a new imaging technique, Harmonic Motion Imaging (HMI), and the evaluation of its potential role in prediction of breast cancer response to neoadjuvant chemotherapy (NACT). The investigators hypothesize that changes in HMI parameters will predict response to neoadjuvant systemic therapy in early-stage breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NACT) is the standard of care for treatment of locally advanced breast cancer (LABC) and inflammatory breast cancer, and is recently being used in earlier stage breast cancer. The ideal outcome of NACT is pathological complete response (pCR), which itself has shown to be associated with improved disease-free survival. However, pCR is currently determined at the time of the surgery when the patient has received the whole cycle of the treatment. Early detection of non-responders to NACT could be used to halt ineffective treatment and start a new chemotherapeutic regimen in order to achieve better tumor response and overall survival. Current techniques to monitor response to NACT based on tumor size changes include mammography, physical examination, ultrasonography and MRI. Clinically assessing tumor size has been shown to be only moderately useful for chemotherapy response prediction in these patients because tumor shrinkage is a late marker of effective treatment. Metabolic activities and microstructure changes induced by NACT can be determined using functional imaging methods such as PET-CT, contrast enhanced MRI and diffuse optical spectroscopy. However, the application of these methods is limited due to high cost and intravenous injection of exogenous contrast agents. Limited studies have shown the potential of ultrasound elastography to be useful in predicting and monitoring response to NACT in breast cancer tumors based on tumor stiffness. Harmonic Motion Imaging (HMI) is a novel ultrasound elastography technique that applies an oscillatory force locally and at different depths in the tissue, in order to determine the characteristics of the resulting localized harmonic motion using high precision tracking methods. Highly localized harmonic motion can be noninvasively generated by ultrasonic beams deep inside the tissue and estimated at high precision, by using RF signals and cross-correlation methods. In addition to not being burdened by the drawbacks encountered by existing techniques, due to the highly localized and harmonic nature of the response, the motion characteristics can be directly linked to the local tissue stiffness. In this study, the investigators propose to compare the changes in the measurements provided by HMI and pathological response rate, between baseline, during treatment and end of the treatment to assess whether HMI can early predict the tumor response to neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥18
* Deemed eligible to receive neoadjuvant systemic therapy as per the treating physician, with the dose and schedule deemed appropriate by the treating physician.
* Any stage invasive breast cancer provided the primary breast tumor size is ≥ 4 mm

Exclusion criteria:

* Patient is pregnant or lactating
* Presence of breast implants
* History of laser or radiation therapy to the affected breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the correlation between change in HMI measurements and pathologic response at completion of neoadjuvant therapy | Baseline and through neoadjuvant therapy completion (an average of 28 weeks)
  * Repeated measures analysis of variance (ANOVA) will be performed to investigate the overall differences in HMI measurements within the tumor and surrounding tissue between responders (pCR and RCB1) and non-responders (RCB2). This relative percent change in tumor stiffness is directly related to HMI measurements.
  * Pathologic response will be assessed by the Residual Cancer Burden (RCB) score, a continuous and categorical measure of pathologic response and an independent predictor of disease free survival. Pathologic response will be dichotomized, with response defined as a score of 0-1 (RCB<2), and no response defined as a score of 2-3 (RCB2).
Assessment of the correlation between change in HMI measurements and pathologic response during neoadjuvant systemic therapy | Baseline and during short-interval on treatment (approximately 4 weeks after treatment initiation)
  * Repeated measures analysis of variance (ANOVA) will be performed to investigate the overall differences in HMI measurements within the tumor and surrounding tissue between responders (pCR and RCB1) and non-responders (RCB2). This relative percent change in tumor stiffness is directly related to HMI measurements.
  * Pathologic response will be assessed by the Residual Cancer Burden (RCB) score, a continuous and categorical measure of pathologic response and an independent predictor of disease free survival. Pathologic response will be dichotomized, with response defined as a score of 0-1 (RCB<2), and no response defined as a score of 2-3 (RCB2).

SECONDARY OUTCOMES:
Assessment of correlation between percent change of tumor size on breast ultrasound and pathologic response at treatment completion | Baseline and through neoadjuvant therapy completion (an average of 28 weeks)
  The investigator will use the statistic Z=(f1-f2)/se where fi= .5ln[(1+ri)/(1-ri)](Fisher transformation of ri), ri is the sample correlation coefficient of Ri and se is the standard error of f1-f2. The investigator will compare Z with standard normal distribution.
Assessment of correlation between percent change of tumor size on breast ultrasound during treatment | Baseline and during short-interval on treatment (approximately 4 weeks after treatment initiation)
  The investigator will use the statistic Z=(f1-f2)/se where fi= .5ln[(1+ri)/(1-ri)](Fisher transformation of ri), ri is the sample correlation coefficient of Ri and se is the standard error of f1-f2. The investigator will compare Z with standard normal distribution.

OTHER OUTCOMES:
Assessment of correlation between change in Ki-67 and change in HMI | Baseline and through neoadjuvant therapy completion (an average of 28 weeks)
  This will be analyzed using Fisher transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Konofagou, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers.

REFERENCES:
- [Background] Saharkhiz N, Ha R, Taback B, Li XJ, Weber R, Nabavizadeh A, Lee SA, Hibshoosh H, Gatti V, Kamimura HAS, Konofagou EE. Harmonic motion imaging of human breast masses: an in vivo clinical feasibility. Sci Rep. 2020 Sep 17;10(1):15254. doi: 10.1038/s41598-020-71960-5. PMID 32943648
- [Background] Hossain MM, Saharkhiz N, Konofagou EE. Feasibility of Harmonic Motion Imaging Using a Single Transducer: In Vivo Imaging of Breast Cancer in a Mouse Model and Human Subjects. IEEE Trans Med Imaging. 2021 May;40(5):1390-1404. doi: 10.1109/TMI.2021.3055779. Epub 2021 Apr 30. PMID 33523806
- [Background] Meng W, Zhang G, Wu C, Wu G, Song Y, Lu Z. Preliminary results of acoustic radiation force impulse (ARFI) ultrasound imaging of breast lesions. Ultrasound Med Biol. 2011 Sep;37(9):1436-43. doi: 10.1016/j.ultrasmedbio.2011.05.022. Epub 2011 Jul 20. PMID 21767903
- See also: Ultrasound Elasticity Imaging Laboratory - Columbia University — https://ueil.bme.columbia.edu/